CLINICAL TRIAL: NCT03643588
Title: Safety and Effectiveness of HYAJOINT Plus Synovial Fluid Supplement for the Treatment of Knee Osteoarthritis Pain
Brief Title: The Comparison of HYAJOINT Plus and Hyalgan Hyaluronan Supplement for Knee Osteoarthritis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDCT-CHP
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Hyaluronan; synovial fluid supplement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYAJOINT Plus group (Experimental): The HYAJOINT Plus group received one intraarticular injection of 3 ml HYAJOINT Plus and be followed for 52 weeks. A single injection of HYAJOINT Plus was performed if criteria was met at 52 weeks, and a 4-weeks follow-up of adverse events was conducted.
  Interventions: Device: HYAJOINT Plus
- Hyalgan group (Active Comparator): The Hyalgan group received intraarticular injection of 2 ml Hyalgan for three continuously weeks and be followed for 52 weeks. A single injection of HYAJOINT Plus was performed if criteria was met at 52 weeks, and a 4-weeks follow-up of adverse events was conducted.
  Interventions: Device: Hyalgan

INTERVENTIONS:
Device: HYAJOINT Plus — Single-injection, 60 mg / 3 ml (2%) cross-linked hyaluronan
  Arms: HYAJOINT Plus group
Device: Hyalgan — Three-injection, 20 mg / 2 ml (1%) linear hyaluronan
  Arms: Hyalgan group

SUMMARY:
The aim of this study was to compare single injection HYAJOINT Plus Synovial Fluid Supplement used on the single and repeat treatment of knee osteoarthritis that has the same safety and effectiveness as three-injection hyaluronan, Hyalgan.

DETAILED DESCRIPTION:
The study was a random, evaluator-blinded, controlled, single center clinical trial. Recruiting patients who have been suffered from the osteoarthritis pain under conventional nonpharmacologic therapy or analgesics for a long time and randomly divided into two groups, HYAJOINT Plus or Hyalgan group, when the inclusion criteria was met and the inform consent was obtained. They were followed for 56 weeks including visits at 4, 12, 26, 39, and 52 weeks post-treatment for the safety and effectiveness evaluation. After complete 52-week visit, subjects would received HYAJOINT Plus on the target knee. These subjects were followed for 4 weeks to assess the safety of repeat treatment or cross reactions of the use from three-injections to single-injection hyaluronan treatment. The primary endpoints were the incidence of any adverse events during the study, as well as the objective assessment of pain visual analog scale at baseline and every visit.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee osteoarthritis for at least 6 months despite nonoperative treatment and/or physical therapy
* Average knee pain score ≧ 30 mm on a 100-mm VAS
* Kellgren-Lawrence grade 2 or 3 knee osteoarthritis based on radiographs taken within previous 6 months 18
* If the VAS pain score of the contralateral knee with radiographic evidence of bilateral knee osteoarthritis was < 30 mm

Exclusion Criteria:

* Hip OA
* Kellgren-Lawrence grade 4 on target knee
* Clinical apparent active symptoms like infections
* Intra-articular injections of hyaluronan within the past 6 months
* Previous orthopaedic surgery on spine or lower limb
* Intra-articular injections of steroid type drugs within the past 3 months
* Diagnosed as Lupus erythematosus, Rheumatoid arthritis, Hemiparesis, Neoplasm or received hemodialysis
* Known allergy to avian proteins or hyaluronic acid products
* Women ascertained or suspected pregnancy or lactating

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
VAS pain score | Baseline, 1, 3, 6, 9 and 12 months post-injection
  The change from baseline in a Visual analog scale score for pain. The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'.
The reported adverse events | 1, 3, 6, 9 and 12 months post-injection
  Any adverse events reported by the patients during the study period and physical examination findings by the evaluator after injections and at each follow-up visit.

SECONDARY OUTCOMES:
WOMAC, Likert Scale | Baseline, 1, 3, 6, 9 and 12 months post-injection
  a 24-item questionnaire with 3 subscales measuring pain, stiffness, and physical function. Total score is 96 and lower scores indicate better outcomes.
VAS stiffness score | Baseline, 1, 3, 6, 9 and 12 months post-injection
  The change from baseline in the Visual analog scale score for stiffness. The VAS scale uses a 100 mm line labelled at '0' with 'no stiffness' and '100' with 'worst stiffness'.
Timed Up-and-Go test (TUG) | Baseline, 1, 3, 6, 9 and 12 months post-injection
  A simple measurement of time in seconds for a subject to rise from an armchair, walk 3 meters, turn around, walk back to the chair, and sit down.
VAS satisfaction score | 1, 3, 6, 9 and 12 months post-injection
  Patients rate their treatment satisfaction based on a 100 mm VAS. The VAS scale uses a 100 mm line labelled at '0' with 'least satisfaction' and '100' with 'highest satisfaction'.

REFERENCES:
- [Derived] Huang TL, Tsai CH. Safety and efficacy of single CHAP Hyaluronan injection versus three injections of linear Hyaluronan in pain relief for knee osteoarthritis: a prospective, 52-week follow-up, randomized, evaluator-blinded study. BMC Musculoskelet Disord. 2021 Jun 23;22(1):572. doi: 10.1186/s12891-021-04467-3. PMID 34162365